CLINICAL TRIAL: NCT00064025
Title: A Phase II Pilot Investigation Of The Relationship Of Short Term Depo-Provera (Medroxyprogesterone Acetate) Exposure To The Morphologic , Biochemical, And Molecular Changes In Primary Endometroid Adenocarcinoma of the Uterine Corpus
Brief Title: Medroxyprogesterone in Treating Patients With Endometrioid Adenocarcinoma of the Uterine Corpus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0211; NCI-2012-02539 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000306440; GOG-0211 (Other: Gynecologic Oncology Group); GOG-0211 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-03

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Adenosquamous Carcinoma; Endometrial Endometrioid Adenocarcinoma, Variant With Squamous Differentiation; Recurrent Uterine Corpus Carcinoma; Stage I Uterine Corpus Cancer; Stage II Uterine Corpus Cancer; Stage III Uterine Corpus Cancer; Stage IV Uterine Corpus Cancer
MeSH Terms: interventions — Medroxyprogesterone; Medroxyprogesterone Acetate

ARMS (1):
- Treatment (medroxyprogesterone) (Experimental): Patients receive medroxyprogesterone intramuscularly once approximately 3 weeks before surgical hysterectomy.
  A subset of 15 patients has tissue collected by pipelle biopsy or curettage at baseline, 72 hours after medroxyprogesterone therapy, and during surgery for gene expression arrays.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Medroxyprogesterone; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Medroxyprogesterone — Given IM
  Other Names: Curretab
Procedure: Therapeutic Conventional Surgery — Undergo surgical hysterectomy

SUMMARY:
This phase II trial is studying how well medroxyprogesterone works in treating patients with endometrioid adenocarcinoma (cancer) of the uterine corpus (the body of the uterus, not including the cervix). Hormone therapy using medroxyprogesterone may be effective in treating endometrioid cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the efficacy of medroxyprogesterone, in terms of induction of histologic response, in patients with progesterone receptor-positive vs progesterone receptor-negative endometrioid adenocarcinoma of the uterine corpus.

II. Determine the early and late changes in gene expression at 72 hours and 21 days in patients treated with this drug.

III. Examine the mechanisms surrounding the dynamic changes in endometrial tumor cells by determining possible correlations among histologic response, steroid receptor status, immunohistochemical measures of growth and apoptosis, and gene expression profiles in patients treated with this drug.

OUTLINE: This is a pilot, multicenter study.

Patients receive medroxyprogesterone intramuscularly once approximately 3 weeks before surgical hysterectomy.

A subset of 15 patients has tissue collected by pipelle biopsy or curettage at baseline, 72 hours after medroxyprogesterone therapy, and during surgery for gene expression arrays.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary endometrioid adenocarcinoma of the uterine corpus

  * All histologic grades and stages eligible
  * Diagnosis by endometrial curettage or biopsy within the past 8 weeks

    * Must have the initial tissue block or 16 unstained sections of 5 micron thickness available
* Performance status - GOG 0-3
* No history of thrombophlebitis or thromboembolic disorders
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No prior therapeutic progesterone or anti-estrogen therapy within 3 months before diagnosis
* No concurrent aminoglutethimide
* No prior cancer treatment that would preclude study therapy
* No concurrent bosentan
* No concurrent rifampin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-04; Primary Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Zaino, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 4/12/2004 and closed to accrual on 9/2/2008.
Groups:
- Depo-Provera: Depo-Provera (Medroxyprogesterone Acetate) 400 mg IM, Given Once, 21-24 Days Prior to Hysterectomy
Period: Overall Study
Arm/Group | Depo-Provera
Started | 75
Completed | 68
Not Completed | 7
Not completed — Ineligible | 4
Not completed — Inevaluable | 3

BASELINE CHARACTERISTICS:
Arm/Group | Depo-Provera
Number analyzed (Participants) | 68
Age, Customized [Number; unit: participants]
  30-39 years | 1
  40-49 years | 3
  50-59 years | 28
  60-69 years | 30
  70-79 years | 3
  80-89 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Histologic Response in Endometrial Adenocarcinomas of the Uterine Corpus That Are Progesterone Receptor Positive Compared With Those That Are Progesterone Receptor Negative
Description: To determine the presence of a histologic response, the slide from the initial sample was compared to the slide from the matching hysterectomy specimen. A complete histologic response was defined as the absence of identifiable adenocarcinoma in the hysterectomy specimen section. A partial histologic response was subjectively defined in advance of the study based on criteria slightly modified from Wheeler et al. (Am J Surg Pathol 2007;31:988-98) as the presence of a complex proliferation of glands that retain the architectural characteristics of adenocarcinoma, but with features of secretion, decreased nuclear stratification, or the presence of eosinophilic, squamous or mucinous metaplasia, when this was absent in the initial sample. A complete or partial histologic response was considered a histologic response in the analysis of data.
  PR Positivity is based on aggregate score >0.2 (vs. <=0.2). Aggregate score based on product of staining intensity and area.
Time Frame: During the hysterectomy, which is 21-24 days after administration of depo-provera
Population: Eligible and Evaluable Patients (patients who had both an intake biopsy and hysterectomy and had histologic response data)
Measure: Number; unit: percentage of participants
Arm/Group | PR Negative (<=0.2) | PR Positive (>0.2)
Number analyzed (Participants) | 8 | 45
percentage of participants | 62.5 | 68.9
Statistical Analysis 1: Comparison: PR Negative (<=0.2) vs PR Positive (>0.2); Test type: Superiority or Other; p = 0.701, Fisher Exact

2. Secondary Outcome: Change From Pre- to Post-treatment in Estrogren Receptor (ER) Expression
Description: Expression is based on an aggregate score based on immunohistochemistry. Staining intensity was scored 1, 2, or 3; and staining area was scored as a percentage (0-100%). The aggregate score is the product of staining intensity and area and ranges from 0 to 3.
Time Frame: During the hysterectomy, which is 21-24 days after administration of depo-provera
Population: Eligible and Evaluable Patients (patients who had both an intake biopsy and hysterectomy)
Measure: Mean (Standard Error); unit: Aggregate Score from Immunohistochemistr
Arm/Group | Depo-Provera
Number analyzed (Participants) | 53
Aggregate Score from Immunohistochemistr | -0.77 (0.14)
Statistical Analysis 1: Comparison: Depo-Provera; Test type: Superiority or Other; p < .001, Paired t-test

3. Secondary Outcome: Change From Pre- to Post-treatment in Progestrogren Receptor (PR) Expression
Description: as for outcome 2
Time Frame: During the hysterectomy , which is 21-24 days after administration of depo-provera
Population: Eligible and Evaluable Patients (patients who had both an intake biopsy and hysterectomy)
Measure: Mean (Standard Error); unit: Aggregate Score from Immunohistochemistr
Arm/Group | Depo-Provera
Number analyzed (Participants) | 53
Aggregate Score from Immunohistochemistr | -1.12 (0.15)
Statistical Analysis 1: Comparison: Depo-Provera; Test type: Superiority or Other; p < .001, Paired t-test

ADVERSE EVENTS:
Time Frame: Toxicity was assessed from the time of study drug administration to the time of the hysterectomy, which occurred 21-24 days after study drug administration.
Description: This study had no Serious Adverse Events (SAEs).
Arm/Group | Depo-Provera
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 39/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Depo-Provera (N=68)
Allergy/Immunology - Other (Immune system disorders) | 1
Leukocytes (Blood and lymphatic system disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 14
Fever (General disorders) | 1
Rigors/Chills (General disorders) | 1
Fatigue (General disorders) | 6
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hot Flashes (Endocrine disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 2
Hemorrhage, Gu - Vagina (Vascular disorders) | 7
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 1
Lymphatics - Other (Blood and lymphatic system disorders) | 2
Edema: Limb (Blood and lymphatic system disorders) | 2
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 1
Bilirubin (Metabolism and nutrition disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 2
Mood Alteration - Depression (Nervous system disorders) | 2
Mood Alteration - Anxiety (Nervous system disorders) | 4
Pain - Other (General disorders) | 1
Pain: Breast (General disorders) | 2
Pain: Uterus (General disorders) | 1
Pain: Head/Headache (General disorders) | 2
Pain: Extremity-Limb (General disorders) | 6
Pain: Rectum (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Urinary Retention (Renal and urinary disorders) | 1
Breast Function (Reproductive system and breast disorders) | 1
Libido (Reproductive system and breast disorders) | 1
Irregular Menses (Reproductive system and breast disorders) | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No